CLINICAL TRIAL: NCT01383291
Title: Postoperative Comparison Between Posterior Prolift Mesh Placement and Posterior IVS Sling Placement
Brief Title: Prolift Versus IVS for Pelvic Floor Prolapse
Status: Withdrawn | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Dr. Menahem Neuman, Western Galilee Hospital and vaious clinics
Other Study IDs: 920090041
Record Dates: First submitted 2011-06-26; First posted 2011-06-28 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Pelvic Floor Prolapse
Keywords: pelvic floor prolapse; prolift; IVS; Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pelvic floor prolapse: Those who underwent prolift and those who underwent IVS

SUMMARY:
* Women who underwent mesh or sling procedures to correct pelvic organ prolapse will be enrolled.
* Their data will be collected from the files.
* Comparison between two groups will be carried our: Those who underwent a posterior IVS and those who underwent posterior prolift procedure.
* The data will be obtained by questionaires by a telephone interview by a physician who did not participate in the surgery.
* Follow-up physical examination data will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Women who previously underwent surgery for pelvic floor prolapse at least a year before

Exclusion Criteria:

* Women who did not have surgery for pelvic floor prolapse

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with pelvic floor prolapse
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2013-01 (Estimated); Study Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Department of Obstetrics and Gynecology, Western Galilee Hospital, Nahariya
  - Clinics of Dr Neuman, Rishon LeZiyyon